CLINICAL TRIAL: NCT00873574
Title: Molecular Study of Factors Involved in JAK-STAT Signalling Pathway in Familial Myeloproliferative Disorders
Brief Title: JAK-STAT Signalling Pathway in Familial Myeloproliferative Disorders
Acronym: SMP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 07014
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Myeloproliferative Disorders
Keywords: Familial myeloproliferative disorders; JAK-STAT; V617; JAK2
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood samples (35 ml) and buccal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 2 patients with MPD for each family. One case for each family will be randomised ; the cohort will be of 120 patients.
  Interventions: Biological: Blood samples and buccal swabs
- 2: 1 control for each family
  Interventions: Biological: Blood samples and buccal swabs

INTERVENTIONS:
Biological: Blood samples and buccal swabs — Peripheral blood samples (35 ml) and buccal swabs

SUMMARY:
The main goal of the study is to progress in our understanding of the molecular basis of myeloproliferative disorders of the bone marrow (polycythemia vera, essential thrombocythemia, primary myelofibrosis). The study will focus on the genes encoding factors implicated in the JAK-STAT pathway which has an essential role in these diseases

DETAILED DESCRIPTION:
Myeloproliferative disorders (MPD) are rare malignant diseases of the bone marrow characterized by a proliferation of differentiated blood cells during a long time and a possible transformation in an acute leukaemia.

The recent identification of a recurrent activating tyrosine kinase mutation V617F in the JAK2 gene provides a breakthrough in the understanding of the molecular mechanisms of these diseases. It can't explain nevertheless the phenotypic diversity of MPD and the occurrence of familial aggregations. The investigators have shown actually that the mutation V617F is a somatic one which is variably expressed among patients in the same family.Other somatic mutations and inherited factors, still unknown, may explain these discrepancies. JAK-STAT pathway has an essential role in non-CML MPD as was shown by the functional consequences of the V617F JAK2 mutation. Therefore, the investigators will focus our study on the genes encoding factors implicated in this signalling pathway. Two genetic approaches will be used: 1-study of known polymorphisms (SNP) of theses genes involved in the JAK-STAT pathway; 2-search of rare mutations located in specific regions (binding domain…) of candidate genes.The study is a national multicenter research based on the national network (55 centers) that the investigators have organized with the help of the French Society Of Hematology in 1998. The investigators propose to include 120 families defined by the presence of at least 2 cases of non CML MPD (WHO and PVSG criteria).The investigators have already collected 60 families (affected cases and control subject); the other 60 will be included in the next two years. In each family, only the two patients with MPD and one control will be included ( all the subjects above 18 years old). Peripheral blood samples (35ml) and buccal swabs will be collected for each subject. Hematologists and ONCOGENETICIANS will include the families, collect all the clinical and biological data and perform the collection of biological material from each subject included in the study according to approved rules.All the data will be anonymously registered on Access data base. Hematological studies will be done in the Immuno-Hematological Laboratory in Saint ANTOINE. Genetic studies will be conducted in the Genetic Department of Saint ANTOINE Hospital now transferred to Pitie-Salpetriere Hospital in Paris. The genetic study will be based on the analysis of 120 unrelated familial SMP cases (randomised) and 120 controls. The investigators will study 10 genes involved in the JAK-STAT pathway ( cytokine receptors, Janus kinases, regulatory factors).The genotyping of SNPs, selected from HAPMAP and CGEMS databases will be performed by quantitative PCR. The investigators plan to analyze 50 SNPs per subject i.e. 24000 genotypes (duplicate points). The analysis will be based on the allelic frequency comparison in the two groups using a bilateral paired t-test; 120 pairs of subjects (case control) allow to detect a 0.6 deviation standard of allelic frequency between cases and controls (alpha = 5%, beta = 10%). The search for rare mutations will be done by genomic sequencing of particular regions in candidates genes in the 120 affected cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected with polycythemia vera, essential thrombocythemia or primary myelofibrosis
* Familial cases
* Subjects above 18 years old
* Non affected controls

Exclusion Criteria:

* patients with chronic myeloid leukaemia
* subjects under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population of familial patients with MPD and controls
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Allelic frequency comparison between the 2 cohorts | At the inclusion visit

SECONDARY OUTCOMES:
Undescribed gene mutations. | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Albert NAJMAN, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Department of Hematology, Hospital Saint Antoine, Paris, France